CLINICAL TRIAL: NCT06750172
Title: Consistency of 24-hour Urinary Aldosterone on on the Second Day and the Third Day in Diagnosis of Primary Aldosteronism Measured in the Oral Sodium Loading Test by Liquid Chromatography-tandem Mass Spectrometry
Brief Title: Simplification of Oral Sodium Loading Test in the Diagnosis of Primary Aldosteronism: 2-day Replacing 3-day Method
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: pumch-06086-08
Record Dates: First submitted 2024-12-06; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Primary Aldosteronism
Keywords: diagnose; the oral sodium loading test
MeSH Terms: conditions — Hyperaldosteronism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma and complete blood cell. 24-hour urine, etc
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary aldosteronism(PA): Inclusion criteria:
  Patients with hypertension and hypokalemia who have been diagnosed with primary aldosteronism following the latest version international guidelines for primary aldosteronism.
  Exclusion criteria:
  * Other causes of endocrine hypertension including pheochromocytoma, Cushing syndrome, etc.
  * Renal artery stenosis and low potassium due to other factors, such as renal tubular acidosis, Bartter syndrome, Gitelman syndrome, etc.
  * History of hyperthyroidism, hepatic and renal insufficiency, malignant tumors, metabolic diseases, cardiovascular diseases, and mental diseases,menstrual disorders
  * Special drugs such as glucocorticoids, immunosuppressants, and oral contraceptives should
  * Diabetes mellitus with HbA1c>7.0% or with insulin or SGLT2 inhibitors were also excluded.
  Interventions: Diagnostic Test: The oral sodium loading test
- healthy control: Inclusion criteria:
  * Age: 20-70 years old, male and female;
  * BMI: 18.5-23.9 kg/m2;
  * Blood pressure: 90-120/60-80 mmHg on three consecutive office blood pressure readings;
  * Female must have regular menstrual cycle (blood and urine samples should be ▪taken during the non-menstrual period);
  * Regular dietary habits;
  * No medications taken within the past 1 month.
  Exclusion criteria:
  History of hypokalemia. History of liver and kidney dysfunction, malignant tumors, metabolic disorders, cardiovascular diseases, and psychiatric disorders, etc.
  Menstrual irregularities and taking contraceptive pills.
  * History of hypertension
  * Have taken any drugs including anti-inflammatory drugs, potassium diuretics, or special health products in the 4 weeks prior to the examination,
  Interventions: Diagnostic Test: The oral sodium loading test

INTERVENTIONS:
Diagnostic Test: The oral sodium loading test — The subjects underwent an oral high-salt diet test with an additional 10g of salt per day for 3 consecutive days, and 24-hour urine measurements of aldosterone, sodium, potassium and creatinine were obtained on days 2 and 3

SUMMARY:
To compare the consistency of 24-hour urinary aldosterone in the diagnosis of primary aldosteronism by oral sodium loading test between the second day method and the third day method

DETAILED DESCRIPTION:
This is an exploratory and prospective study of 17 healthy controls and 15 patients with primary aldosteronism, in which each participant will receive a high-sodium diet for 3 days to conduct a confirmatory test for primary aldosteronism. The consistency between the 2-day and 3-day oral sodium loading test for the diagnosis of primary aldosteronism is compared by measuring the 24-hour urinary aldosterone levels of the participants on the second and third days of the high-sodium diet. The study aims to explore whether the 24-hour urinary aldosterone level on the second day can replace the 24-hour urinary aldosterone level on the third day for the diagnosis of primary aldosteronism.

ELIGIBILITY:
PA patients:

Inclusion criteria:

* Patients with hypertension and hypokalemia who have been diagnosed with primary aldosteronism following the latest version international guidelines for primary aldosteronism.
* Age: 20-70 years old, male and female;
* BMI: 18.5-23.9 kg/m2;

Exclusion criteria:

* Other causes of endocrine hypertension including pheochromocytoma, Cushing syndrome, etc.
* Renal artery stenosis and low potassium due to other factors, such as renal tubular acidosis, Bartter syndrome, Gitelman syndrome, etc.
* History of hyperthyroidism, hepatic and renal insufficiency, malignant tumors, metabolic diseases, cardiovascular diseases, and mental diseases,menstrual disorders Healthy volunteers

Inclusion criteria:

* Age: 20-70 years old, male and female;
* BMI: 18.5-23.9 kg/m2;
* Blood pressure: 90-120/60-80 mmHg on three consecutive office blood pressure readings;
* Female must have regular menstrual cycle (blood and urine samples should be taken during the non-menstrual period);
* Regular dietary habits;
* No medications taken within the past 1 month.

Exclusion criteria:

* History of hypokalemia.
* History of liver and kidney dysfunction, malignant tumors, metabolic disorders, cardiovascular diseases, and psychiatric disorders, etc.
* Menstrual irregularities and taking contraceptive pills.
* History of hypertension
* Have taken any drugs including anti-inflammatory drugs, potassium diuretics, or special health products in the 4 weeks prior to the examination,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers and patients with primary aldosteronism in a single tertiary hospital center
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Consistency of 2-day and 3-day 24h urinary aldosterone in the oral sodium load test | 4 day
  To explore whether there was statistical difference in the 24h urinary aldosterone on the 2nd day and the 3rd day detected by LC-MS (Liquid chromatography-tandem mass spectrometry) in oral sodium load test, and to study whether the 2-day method can replace the 3-day method in the diagnosis of primary aldosteronism

SECONDARY OUTCOMES:
Consistency of 2-day and 3-day PAC(Plasma aldosterone concentration) in the oral sodium load test | 4 day
  To explore whether there was statistical difference in plasma aldosterone concentration on the second day and the third day in oral sodium load test, and to study whether the 2-day method can replace the 3-day method in the diagnosis of primary aldosteronism.
Consistency of the plasma renin activity on the second day and the third day in oral sodium load test | 4 day
  To explore whether there was statistical difference in the plasma renin activity on the second day and the third day in oral sodium load test, and to study whether the 2-day method can replace the 3-day method in the diagnosis of primary aldosteronism
consistency of the the aldosterone-to-renin ratio(ARR) on the second day and the third day in oral sodium load test | 4 day
  To explore whether there was statistical difference in the aldosterone-to-renin ratio on the second day and the third day in oral sodium load test, and to study whether the 2-day method can replace the 3-day method in the diagnosis of primary aldosteronism

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turcu AF, Yang J, Vaidya A. Primary aldosteronism - a multidimensional syndrome. Nat Rev Endocrinol. 2022 Nov;18(11):665-682. doi: 10.1038/s41574-022-00730-2. Epub 2022 Aug 31. PMID 36045149
- [Background] Funder JW. Sensitivity to aldosterone: plasma levels are not the full story. Hypertension. 2014 Jun;63(6):1168-70. doi: 10.1161/HYPERTENSIONAHA.114.03127. Epub 2014 Apr 7. No abstract available. PMID 24711520
- [Background] Kline GA, Darras P, Leung AA, So B, Chin A, Holmes DT. Surprisingly low aldosterone levels in peripheral veins following intravenous sedation during adrenal vein sampling: implications for the concept of nonsuppressibility in primary aldosteronism. J Hypertens. 2019 Mar;37(3):596-602. doi: 10.1097/HJH.0000000000001905. PMID 30703073
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Background] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310